CLINICAL TRIAL: NCT03782545
Title: Multi-Center Pilot Study of Cutera truSculpt Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cutera Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-18-TS-18
Record Dates: First submitted 2018-12-17; First posted 2018-12-20 (Actual); Results first posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: Treatment for Cellulite on the Stomach and Flanks

STUDY DESIGN:
Intervention Model Description: A type of intervention model describing a clinical trial in which all participants receive the same intervention/treatment.
Masking Description: This is an open label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment with the truSculpt RF device (Experimental): Subjects will be treated with the truSculpt RF device
  Interventions: Device: Cutera truSculpt Device

INTERVENTIONS:
Device: Cutera truSculpt Device — The Cutera truSculpt Device uses radio frequency (RF) energy to provide topical heating for the purpose of elevating tissue temperature for the treatment of selected medical conditions, such as temporary reduction in the appearance of cellulite.

SUMMARY:
Exploratory study to evaluate the safety, efficacy and ergonomics of Cutera truSculpt device.

DETAILED DESCRIPTION:
This study will evaluate the safety, efficacy and ergonomics of Cutera truSculpt device.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subject must be able to read, understand and sign the Informed Consent Form.

  2. Female or Male, 18 to 65 years of age (inclusive). 3. Subject has visible fat bulges in the area to be treated. 4. Non-smoking for at least 6 months and willing to refrain from smoking for the duration of the study.

  5. Subject must agree to not undergo any other procedure(s) in the treatment region during the study period.

  6. Subject must adhere to the follow-up schedule and study instructions. 7. Subject must adhere to the same diet and/or exercise routine throughout the study, and agree to maintain the same weight throughout the study.

  8. Willing to have photographs taken of the treatment area and agree to use of photographs for presentation, (educational and/or marketing), publications, and any additional marketing purposes.

  9. For female subjects: not pregnant or lactating and is either post-menopausal, surgically sterilized, or using a medically acceptable form of birth control prior to enrollment and during the entire course of the study.

Exclusion Criteria:

1. Participation in a clinical trial of another device or drug within 1 month of study participation, or during the study period.
2. Any type of prior cosmetic treatment to the target area within 6 months of study participation.
3. Any prior invasive cosmetic surgery to the target area, such as liposuction.
4. Has a pacemaker, internal defibrillator, implantable cardioverter-defibrillator, nerve stimulator implant, cochlear implant or any other electronically, magnetically or mechanically activated implant.
5. Has metal implant(s) within the body, such as artificial heart valves.
6. Significant uncontrolled concurrent illness that in the opinion of the Investigator would make the subject unsuitable for inclusion.
7. History of any disease or condition that could impair wound healing.
8. History of keloid formation, hypertrophic scarring or abnormal/delayed wound healing.
9. Skin abnormality in the treatment area that in the opinion of the Investigator would make the subject unsuitable for inclusion.
10. Currently undergoing systemic chemotherapy or radiation treatment for cancer, or history of treatment in the target area within 3 months of study participation.
11. Allergy or sensitivity to Tegaderm.
12. As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study or a condition that would compromise the subject's ability to comply with the study requirements.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-05-11 (Actual); Primary Completion 2018-12-19 (Actual); Study Completion 2018-12-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Laser and Skin Surgery Center of Northern California, Sacramento, California
  - Advanced Dermatology, Glencoe, Illinois
  - Union Square Dermatology, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Researchers involved in the study will have access to the final study data.
Supporting Information: Study Protocol, ICF, CSR

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment With the truSculpt RF Device
Started | 34
Completed | 30
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Treatment With the truSculpt RF Device
Number analyzed (Participants) | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 34
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: GAIS at 12 Weeks Post Final Treatment
Description: Global Aesthetic Improvement Scale will be assessed at 12 weeks post final treatment by the investigator by comparing against Baseline photos Higher scores indicate better outcomes 0= No change
  1. Mild Improvement
  2. Moderate improvement
  3. Significant Improvement
Time Frame: 12 weeks post final treatment
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Treatment With the truSculpt RF Device
Number analyzed (Participants) | 30
score on a scale | 2 (0.94)

ADVERSE EVENTS:
Time Frame: up to 12 weeks post final treatment
Arm/Group | Treatment With the truSculpt RF Device
All-Cause Mortality (participants affected / at risk) | 0/34
Serious Adverse Events (participants affected / at risk) | 0/34
Other Adverse Events (participants affected / at risk) | 22/34
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment With the truSculpt RF Device (N=34)
Erythema (Skin and subcutaneous tissue disorders) | 22
Edema (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2018-04-26): https://cdn.clinicaltrials.gov/large-docs/45/NCT03782545/Prot_001.pdf